CLINICAL TRIAL: NCT04999982
Title: Pilot Testing PRE-CARE to Address Unmet Social Needs for Preschoolers With Inattention and/or Hyperactivity
Brief Title: Pilot Testing PREschooler Care, Community Resources, Advocacy, Referral, Education (PRE-CARE)
Acronym: PRE-CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Andrea Spencer, Vice Chair for Research, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 2023-6209; 5K23MH118478-03 (NIH)
Record Dates: First submitted 2021-08-03; First posted 2021-08-11 (Actual); Results first posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Attention Deficit/Hyperactivity Disorder; Inattention
Keywords: Parent; Caregiver; Community health worker
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group- PRE-CARE (Experimental): Participants will receive the 1:1 PRE-CARE social needs navigation intervention with specific content and delivery strategy which was developed based on 1) quantitative analyses of the association between unmet social needs and ADHD symptoms in a large-scale nationally representative sample of children age 3-5, and 2) in-depth qualitative interviews with parents/guardians of preschoolers with inattention and/or hyperactivity symptoms to identify mechanisms by which unmet social needs exacerbate ADHD symptoms and functioning.
  Interventions: Other: Screening; Other: Resource Packet; Other: Resource Navigation
- Control group- Care as Usual (Active Comparator): Families randomly assigned to the control condition will continue to receive care as usual, which includes screening for social needs annually at well-child visits as recommended by the American Academy of Pediatrics (AAP), followed by provision of information as needed by the family. Families will also be offered the opportunity to make research assessments available to their primary care physician for best continuity of care.
  Interventions: Other: Care as usual

INTERVENTIONS:
Other: Screening — Parent-report screening for remediable, unmet social needs.
  Arms: Intervention group- PRE-CARE
Other: Resource Packet — Provision of packet of resource sheets ("Family Resource Booklet") detailing local community-based resources to address these needs, with needs that respond to family's requests highlighted.
  Arms: Intervention group- PRE-CARE
Other: Resource Navigation — Navigation to resources, care coordination, and parent support provided by a trained bachelors-level interventionist.
  Arms: Intervention group- PRE-CARE
Other: Care as usual — Screening for social needs annually at well-child visits as recommended by the AAP followed by provision of information as needed by the family.
  Arms: Control group- Care as Usual

SUMMARY:
The goal of this proposed study is to pilot test a novel treatment model (PRE-CARE) addressing unmet social needs for families of preschool-age children with Attention Deficit/Hyperactivity Disorder (ADHD) symptoms. The investigators will conduct an adaptive, pilot randomized controlled trial (RCT) of the intervention with parents of 60 low-income children age 3-5 (36-71 months) with ADHD symptoms in order to: optimize intervention delivery; field test study logistics (e.g., recruitment, enrollment, randomization, retention); explore putative intervention mechanisms; and obtain estimates of study parameters to plan an appropriately powered RCT of the intervention.

The PRE-CARE intervention is adapted from Well Child Care, Evaluation, Community, Resources, Advocacy, Referral, Education (WE CARE), a screening and referral intervention that has been shown to be feasible and effective in addressing the family psychosocial stressors of low-income families seen in pediatric medical homes. Given the negative impact that socioeconomic stressors can have on the health and development of young children with ADHD symptoms, tailored interventions such as PRE-CARE may serve as a vital early intervention strategy to promote long-term well-being.

ELIGIBILITY:
Inclusion Criteria:

* Legal guardian and primary caregiver of a child aged 36-71 months
* Legal guardian or primary caregiver is age 16 years or older
* Child receives pediatric care at Boston Medical Center or at one of the participating affiliated clinics
* Able to understand informed consent procedures in English or Spanish
* Participant has a child aged 36-71 months with an ADHD diagnosis, OR one elevated total or subscale score at the 80th percentile on the ADHD-Rating Scale-IV Preschool Version. 80th percentile cut-offs on the ADHD-Rating Scale-IV Preschool Version are as follows:

  * For male children, a total score ≥ 25 OR subscale score (inattention and/or hyperactivity) ≥ 12
  * For female children, a total score ≥ 13 OR subscale score (inattention and/or hyperactivity) ≥ 6 for female children

Exclusion Criteria:

* There are no specific exclusion criteria for this study

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2025-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Spencer, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (2):
- United States (2):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We enrolled 54 parents but only 45 parents were ultimately randomized, hence the discrepancy between enrollment and participant flow.
Period: Overall Study
Arm/Group | Intervention Group- PRE-CARE | Control Group- Care as Usual
Started | 22 | 23
Completed | 16 | 17
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group- PRE-CARE | Control Group- Care as Usual | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 23 | 45
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 35.0 [33.0 to 40.0] | 32.0 [27.5 to 35.0] | 34.0 [30.0 to 64.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 10 | 10 | 20
  Non-Hispanic Black | 7 | 8 | 15
  Non-Hispanic White | 2 | 4 | 6
  More than one race | 2 | 1 | 3
  Other race | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 23 | 45

OUTCOME MEASURES:

1. Primary Outcome: ADHD Symptoms
Description: ADHD-Rating Scale (RS)-IV Preschool Version is a parent-report survey that measures presence and severity of ADHD symptoms for preschoolers. In our study, we used this measure to assess overall ADHD symptom burden. The 18-item validated scale asks parents about the 18 diagnostic criteria for ADHD and how often their child exhibits each symptom. The scale can be used as an overall score (total symptoms) or by subscales (9-item inattention subscale and 9-item hyperactivity subscale). Responses are reported by parents for each item along a 4-point Likert scale from 0 to 3, where 0=rarely or never and 3=very often. For our purposes, we computer the total score for a measure of total ADHD symptom severity, and did not use the subscales. Total scores range from 0 to 54, where lower is less ADHD symptoms/lower symptom severity, and higher scores represent higher symptom severity.
Time Frame: Baseline, 3 months, 6 months, and 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group- PRE-CARE | Control Group- Care as Usual
Number analyzed (Participants) | 22 | 23
score on a scale
  Baseline | 27.7 (15.5) | 27.5 (14.4)
  3 months | 27.7 (17.9) | 34.6 (14.2)
  6 months | 21.5 (15.2) | 27.6 (16.7)
  12 months | 21.0 (16.8) | 23.8 (16.5)

2. Primary Outcome: Total Resources Enrolled (Parent Report)
Description: Resource access was measured based on a parent report checklist of resources enrolled. The checklist was based on the Child HealthWatch Survey and modeled after data collected for the clinical trial testing the original social determinants intervention on which this intervention is based. The checklist included 18 resources that families could be enrolled in (for example - healthcare services, mental health care, special education, food benefits, housing assistance, etc), and asked parents to indicate which resources they were enrolled in. The end result is a count between 0 and 18 representing how many resources their family was enrolled in. Higher numbers indicate higher number of resources enrolled, whereas lower numbers indicate lower number of resources enrolled.
Time Frame: Baseline, 3 months, 6 months, 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group- PRE-CARE | Control Group- Care as Usual
Number analyzed (Participants) | 22 | 23
units on a scale
  Baseline | 3.4 (2.3) | 4.1 (2.7)
  3 months | 4.7 (2.7) | 4.1 (2.3)
  6 months | 4.7 (3.1) | 4.1 (2.4)
  12 months | 4.3 (2.5) | 4.6 (2.6)

3. Secondary Outcome: Child Psychiatric Symptoms
Description: The Child Behavior Checklist 1.5-5 (CBCL 1.5/5) is a standardized tool used to assess child psychiatric symptoms for children 1.5-5 years old. The questionnaire obtains caregivers' ratings of 99 problem items along a Likert scale. Parents/caregivers rate each item 0=not true, 1=somewhat or sometimes true, 2=very true or often true of the child (based on the preceding 6 months). Higher scores are correlated with more psychiatric symptoms. Items can be grouped into syndrome scales or the total score can be used to represent overall psychiatric symptom severity. Here we use the total score to represent total psychiatric symptoms. Scores are reported as t-scores, where 50 indicates the population mean with a standard deviation of 10. Higher scores indicate more symptoms. On this scale, scores between 65 and 69 are considered borderline elevated, and scores of 70 or more are considered clinically significant.
Time Frame: Baseline, 6 months, 12 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Intervention Group- PRE-CARE | Control Group- Care as Usual
Number analyzed (Participants) | 22 | 23
T-score
  Baseline | 62.6 (13.8) | 59.0 (15.0)
  6 months | 49.0 (16.0) | 51.0 (19.6)
  12 months | 48.3 (17.2) | 48.1 (18.5)

4. Secondary Outcome: Parental Depression
Description: Patient Health Questionnaire (PHQ)-9 will be used to measure frequency and severity of parental symptoms of depression within the past two weeks. The measure is the major depressive disorder (MDD) module of the full PHQ, and scores each of the 9 Diagnostic and Statistical Manual criteria of MDD as "0" (not at all) to "3" (nearly every day), providing a 0-27 severity score. Higher scores are correlated with more parental depression.
Time Frame: baseline, 3 months, 6 months, 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group- PRE-CARE | Control Group- Care as Usual
Number analyzed (Participants) | 22 | 23
score on a scale
  Baseline | 7.0 (6.7) | 5.7 (5.8)
  3 months | 7.1 (7.5) | 8.8 (8.5)
  6 months | 5.8 (5.3) | 6.3 (6.7)
  12 months | 6.6 (6.1) | 6.9 (7.7)

5. Secondary Outcome: Parental Attention-deficit/Hyperactivity Disorder (ADHD)
Description: Adult ADHD Self-Report Scale (ASRS-v1.1) Symptom Checklist will be used to measure parent ADHD symptoms. The measure consists of 18 items matching Diagnostic and Statistical Manual IV criteria for adult ADHD. Items are scored on a 5-point Likert scale, (Never, Rarely, Sometimes, Often, Very Often). The questionnaire is scored based on number of symptoms, leadng to a score between 0 and 18 for the questionnaire. Items 1, 2, 3, 9, 12, 16, 18 are each counted as a symptom (1 point each) if the participant answers Sometimes, Often, or Very Often. Items 4, 5, 6, 7, 8, 10, 11, 13, 14, 15, 17 are each counted as a symptom (1 point each) if the participant answers Often or Very Often. Higher scores indicate higher symptom burden.
Time Frame: baseline, 3 months, 6 months, 12 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group- PRE-CARE | Control Group- Care as Usual
Number analyzed (Participants) | 22 | 23
score on a scale
  Baseline | 3 [1 to 6] | 3 [0 to 6]
  3 months | 4 [0 to 5] | 3 [0 to 6]
  6 months | 1 [0 to 4] | 1 [0 to 5]
  12 months | 1 [0 to 6] | 0 [0 to 2]

6. Secondary Outcome: Global Perceived Stress
Description: The Perceived Stress Scale (PSS) will be used to measure perceptions of levels of stress within the past month using 10 items on a 4 point Likert scale indicating 0 = Never, 1 = Almost Never, 2 = Sometimes, 3 = Fairly Often, and 4 = Very Often. Higher scores [range 0 to 40] are correlated with more perceived stress.
Time Frame: baseline, 3 months, 6 months, 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group- PRE-CARE | Control Group- Care as Usual
Number analyzed (Participants) | 22 | 23
score on a scale
  Baseline | 17.1 (5.0) | 20.1 (5.4)
  3 Months | 16.1 (5.1) | 20.1 (4.2)
  6 months | 16.5 (7.0) | 20.3 (5.9)
  12 months | 16.1 (5.6) | 19.5 (4.7)

7. Secondary Outcome: Parenting Stress
Description: The Parenting Stress Inventory, Short Form (PSI-4-SF) will be used to measure specific levels of stress in relation to taking care of their child and the parent-child system. The scale includes 36 items, each of which uses a 4-point Likert scale from Strongly Disagree to Strongly Agree. The scale includes subscales and a Total score representing total stress on parents, reported here. Possible scores range from 36 to 180. Higher scores are correlated with more parental stress.
Time Frame: baseline, 3 months, 6 months, 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group- PRE-CARE | Control Group- Care as Usual
Number analyzed (Participants) | 22 | 23
score on a scale
  Baseline | 90.3 (24.6) | 75.6 (30.6)
  3 months | 98.2 (23.8) | 83.4 (22.2)
  6 months | 89.9 (29.8) | 86.5 (17.9)
  12 months | 93.5 (25.1) | 87.1 (22.2)

8. Secondary Outcome: PRE-CARE Feasibility and Acceptability Questionnaire
Description: The PRE-CARE Feasibility and Acceptability Questionnaire will be used to measure intervention satisfaction using 14 items on a 4 point Likert scale. Items will ask about satisfaction of information and resources provided, length of intervention, perceived helpfulness of intervention, and whether or not they would recommend the program to a parent of a similarly aged child. Higher scores are correlate with greater satisfaction.
Time Frame: 3 months
Population: Reporting percent of participants who agreed or strongly disagreed with each item
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group- PRE-CARE
Number analyzed (Participants) | 16
Participants
  PRE-CARE helped me to access resources for my family: Agree/Strongly Agree | 15
  PRE-CARE helped me to access resources for my family: Disagree/Strongly Disagree | 1
  PRE-CARE helped me to access resources for my family: Missing | 0
  PRE-CARE was not necessary for me and my child: Agree/Strongly Agree | 2
  PRE-CARE was not necessary for me and my child: Disagree/Strongly Disagree | 14
  PRE-CARE was not necessary for me and my child: Missing | 0
  I was satisfied with the information provided in the family resource booklet: Agree/Strongly Agree | 16
  I was satisfied with the information provided in the family resource booklet: Disagree/Strongly Disagree | 0
  I was satisfied with the information provided in the family resource booklet: Missing | 0
  I was satisfied with the service provided in PRE-CARE: Agree/Strongly Agree | 16
  I was satisfied with the service provided in PRE-CARE: Disagree/Strongly Disagree | 0
  I was satisfied with the service provided in PRE-CARE: Missing | 0
  I think the family resource booklet was clear and easy to understand: Agree/Strongly Agree | 16
  I think the family resource booklet was clear and easy to understand: Disagree/Strongly Disagree | 0
  I think the family resource booklet was clear and easy to understand: Missing | 0
  I think there was too much information provided: Agree/Strongly Agree | 4
  I think there was too much information provided: Disagree/Strongly Disagree | 12
  I think there was too much information provided: Missing | 0
  I think there was not enough information provided: Agree/Strongly Agree | 5
  I think there was not enough information provided: Disagree/Strongly Disagree | 11
  I think there was not enough information provided: Missing | 0
  I was satisfied with the quality of PRE-CARE: Agree/Strongly Agree | 16
  I was satisfied with the quality of PRE-CARE: Disagree/Strongly Disagree | 0
  I was satisfied with the quality of PRE-CARE: Missing | 0
  I had no difficulty understanding the information provided during PRE-CARE: Agree/Strongly Agree | 15
  I had no difficulty understanding the information provided during PRE-CARE: Disagree/Strongly Disagree | 1
  I had no difficulty understanding the information provided during PRE-CARE: Missing | 0
  PRE-CARE was too short: Agree/Strongly Agree | 7
  PRE-CARE was too short: Disagree/Strongly Disagree | 9
  PRE-CARE was too short: Missing | 0
  PRE-CARE took too much time: Agree/Strongly Agree | 2
  PRE-CARE took too much time: Disagree/Strongly Disagree | 13
  PRE-CARE took too much time: Missing | 1
  The resources I received will not improve my child's health or symptoms: Agree/Strongly Agree | 4
  The resources I received will not improve my child's health or symptoms: Disagree/Strongly Disagree | 12
  The resources I received will not improve my child's health or symptoms: Missing | 0
  I would recommend PRE-CARE to another parent of a preschool-age child: Agree/Strongly Agree | 16
  I would recommend PRE-CARE to another parent of a preschool-age child: Disagree/Strongly Disagree | 0
  I would recommend PRE-CARE to another parent of a preschool-age child: Missing | 0

ADVERSE EVENTS:
Time Frame: Collected for 12 months after enrollment for each subject.
Arm/Group | Intervention Group- PRE-CARE | Control Group- Care as Usual
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT04999982/Prot_SAP_000.pdf